CLINICAL TRIAL: NCT00447330
Title: A Phase ll Study of Oxaliplatin, Capecitabine, and Bevacizumab in the Treatment of Metastatic Esophagogastric Adenocarcinomas
Brief Title: Oxaliplatin, Capecitabine and Avastin for Metastatic Esophagogastric Adenocarcinoma
Acronym: XAGastric
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Hoffmann-La Roche (Industry); Sanofi (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00008710; 11100 (Other: Old FDA IND Number); 8797 (Other: Duke legacy protocol number)
Record Dates: First submitted 2007-03-13; First posted 2007-03-14 (Estimated); Results first posted 2015-01-28 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2014-07

CONDITIONS: Esophageal Neoplasms; Stomach Neoplasms; Neoplasm Metastasis
Keywords: metastatic esophagogastric adenocarcinomas; ESOPHAGEAL CANCER; GASTRIC CANCER; ADENOCARCINOMA; TARGTED THERAPY; BEVACIZUMAB; CAPECITBAINE; OXALIPLATIN; METASTATIC
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Neoplasm Metastasis; Adenocarcinoma | interventions — Capecitabine; Oxaliplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: capecitabine (Xeloda), oxaliplatin and bevacizumab (Avastin)

INTERVENTIONS:
Drug: capecitabine (Xeloda), oxaliplatin and bevacizumab (Avastin) — Capecitabine will be administered orally at a twice daily dose of 850 mg/m2 (equivalent to a total daily dose of 1700 mg/m2) given days 1-14 of the three week cycle.
  Oxaliplatin will be administered at the dose of 130 mg/m2 given as a 2-hour intravenous infusion on day 1 of a three week cycle.
  Bevacizumab will be administered at a dose of 15 mg/kg given as a 30-90 minute intravenous infusion on day 1 of a three week cycle following the administration of oxaliplatin.

SUMMARY:
The purpose of this study is to evaluate the progression free survival of capecitabine (Xeloda), oxaliplatin and bevacizumab (Avastin) in previously untreated metastatic esophagogastric adenocarcinomas.

DETAILED DESCRIPTION:
The number of new cases of esophageal and gastric cancers in the United States in 2005 is 14520 for esophageal cancer and 21860 for gastric cancer. Unfortunately, esophageal and gastric cancers will also account for 13570 and 11550 deaths, respectively, in 2005. The 5 year survival rates for metastatic gastroesophageal, GE junctional, and gastric cancers are less than 5%. The major current treatment modality for patients with advanced esophageal, GE junctional, and gastric adenocarcinomas is systemic chemotherapy.

We seek to investigate the efficacy of capecitabine and oxaliplatin in combination with bevacizumab as first line treatment for metastatic esophagogastric cancers. The choice of capecitabine and oxaliplatin is made to develop a user-friendly biologically-based regimen, offering patients oral capecitabine in place of continuous 5FU infusion pumps. Since capecitabine can be given crushed this regimen may both be active and user-friendly. Preliminary data in colorectal cancer suggest that the regimen of capecitabine, oxaliplatin, and bevacizumab has comparable activity to FOLFOX-bevacizumab. The goal of the proposed regimen is to define a capecitabine and oxaliplatin-based regimen that optimizes biological approaches over cytotoxic approaches. The addition of bevacizumab to chemotherapy regimens for metastatic colorectal cancer, metastatic non-small cell lung cancer, and metastatic breast cancer has shown to improve response rates and overall survival. If active, this regimen could serve as a first line comparator to the capecitabine, oxaliplatin, and epirubicin combination. This approach will also help to simplify regimen development across gastrointestinal cancers.

In addition to the primary efficacy endpoint of this protocol, several correlative endpoints will also be examined in an exploratory manner. The importance of developing blood-based and tumor biomarkers has been extensively reviewed. However, the role of such predictive markers has not been well studied for XELOX-A. This information is important since it may help define which populations are most likely to benefit and most likely to suffer significant toxicity from this important GI cancer regimen. This biomarker approach may also help understand and define mechanisms of sensitivity, resistance, and toxicity that may be used to guide future hypothesis-driven studies designed to improve the efficacy and safety of this regimen. The correlative biomarker endpoints include serum, plasma and urine biomarkers (e.g. VEGF and bFGF), a wound healing model of angiogenesis, and tumor biopsy studies .

ELIGIBILITY:
Primary Inclusion Criteria:

* Histologically or cytologically documented and radiographically measurable adenocarcinoma of the esophagus or stomach that is metastatic/recurrent and not amenable to potentially curative treatment
* No prior therapy for metastatic disease
* Prior radiation therapy is permitted, provided it is completed > 28 days prior to day 1 of study drug
* Normal organ and marrow function
* Karnofsky Performance Status 70-100%

Primary Exclusion Criteria:

* Unstable or poorly controlled hypertension > 150/100 mm Hg
* Arterial thromboembolic events within 6 months
* Clinically significant uncontrolled cardiac disease
* Significant proteinuria at baseline
* Grade 2 or greater peripheral neuropathy
* History of abdominal fistula, GI perforation, or intra-abdominal abscess within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-02; Primary Completion 2014-01 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hope E Uronis, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - University of Wake Forest Baptist Medical Center, Winston-Salem, North Carolina

REFERENCES:
- [Background] Jemal A, Murray T, Ward E, Samuels A, Tiwari RC, Ghafoor A, Feuer EJ, Thun MJ. Cancer statistics, 2005. CA Cancer J Clin. 2005 Jan-Feb;55(1):10-30. doi: 10.3322/canjclin.55.1.10. PMID 15661684
- [Background] Bollschweiler E, Wolfgarten E, Gutschow C, Holscher AH. Demographic variations in the rising incidence of esophageal adenocarcinoma in white males. Cancer. 2001 Aug 1;92(3):549-55. doi: 10.1002/1097-0142(20010801)92:33.0.co;2-l. PMID 11505399
- [Background] Wijnhoven BP, Siersema PD, Hop WC, van Dekken H, Tilanus HW. Adenocarcinomas of the distal oesophagus and gastric cardia are one clinical entity. Rotterdam Oesophageal Tumour Study Group. Br J Surg. 1999 Apr;86(4):529-35. doi: 10.1046/j.1365-2168.1999.01082.x. PMID 10215831
- [Background] Glimelius B, Ekstrom K, Hoffman K, Graf W, Sjoden PO, Haglund U, Svensson C, Enander LK, Linne T, Sellstrom H, Heuman R. Randomized comparison between chemotherapy plus best supportive care with best supportive care in advanced gastric cancer. Ann Oncol. 1997 Feb;8(2):163-8. doi: 10.1023/a:1008243606668. PMID 9093725
- [Background] Hsu CH, Yeh KH, Chen LT, Liu JM, Jan CM, Lin JT, Chen YC, Cheng AL. Weekly 24-hour infusion of high-dose 5-fluorouracil and leucovorin in the treatment of advanced gastric cancers. An effective and low-toxic regimen for patients with poor general condition. Oncology. 1997 Jul-Aug;54(4):275-80. doi: 10.1159/000227702. PMID 9216850
- [Background] Leichman L, McDonald B, Dindogru A, Samson M, Vaitkevicius VK. Cisplatin. An active drug in the treatment of disseminated gastric cancer. Cancer. 1984 Jan 1;53(1):18-22. doi: 10.1002/1097-0142(19840101)53:13.0.co;2-j. PMID 6317158
- [Background] Webb A, Cunningham D, Scarffe JH, Harper P, Norman A, Joffe JK, Hughes M, Mansi J, Findlay M, Hill A, Oates J, Nicolson M, Hickish T, O'Brien M, Iveson T, Watson M, Underhill C, Wardley A, Meehan M. Randomized trial comparing epirubicin, cisplatin, and fluorouracil versus fluorouracil, doxorubicin, and methotrexate in advanced esophagogastric cancer. J Clin Oncol. 1997 Jan;15(1):261-7. doi: 10.1200/JCO.1997.15.1.261. PMID 8996151
- [Background] Miwa M, Ura M, Nishida M, Sawada N, Ishikawa T, Mori K, Shimma N, Umeda I, Ishitsuka H. Design of a novel oral fluoropyrimidine carbamate, capecitabine, which generates 5-fluorouracil selectively in tumours by enzymes concentrated in human liver and cancer tissue. Eur J Cancer. 1998 Jul;34(8):1274-81. doi: 10.1016/s0959-8049(98)00058-6. PMID 9849491
- [Background] Schuller J, Cassidy J, Dumont E, Roos B, Durston S, Banken L, Utoh M, Mori K, Weidekamm E, Reigner B. Preferential activation of capecitabine in tumor following oral administration to colorectal cancer patients. Cancer Chemother Pharmacol. 2000;45(4):291-7. doi: 10.1007/s002800050043. PMID 10755317
- [Background] Hong YS, Song SY, Lee SI, Chung HC, Choi SH, Noh SH, Park JN, Han JY, Kang JH, Lee KS, Cho JY. A phase II trial of capecitabine in previously untreated patients with advanced and/or metastatic gastric cancer. Ann Oncol. 2004 Sep;15(9):1344-7. doi: 10.1093/annonc/mdh343. PMID 15319239
- [Background] Koizumi W, Saigenji K, Ujiie S, Terashima M, Sakata Y, Taguchi T; Clinical Study Group of Capecitabine. A pilot phase II study of capecitabine in advanced or recurrent gastric cancer. Oncology. 2003;64(3):232-6. doi: 10.1159/000069313. PMID 12697963
- [Background] Kim TW, Kang YK, Ahn JH, Chang HM, Yook JH, Oh ST, Kim BS, Lee JS. Phase II study of capecitabine plus cisplatin as first-line chemotherapy in advanced gastric cancer. Ann Oncol. 2002 Dec;13(12):1893-8. doi: 10.1093/annonc/mdf323. PMID 12453857
- [Background] Evans TR, Pentheroudakis G, Paul J, McInnes A, Blackie R, Raby N, Morrison R, Fullarton GM, Soukop M, McDonald AC. A phase I and pharmacokinetic study of capecitabine in combination with epirubicin and cisplatin in patients with inoperable oesophago-gastric adenocarcinoma. Ann Oncol. 2002 Sep;13(9):1469-78. doi: 10.1093/annonc/mdf243. PMID 12196374
- [Background] Al-Batran SE, Atmaca A, Hegewisch-Becker S, Jaeger D, Hahnfeld S, Rummel MJ, Seipelt G, Rost A, Orth J, Knuth A, Jaeger E. Phase II trial of biweekly infusional fluorouracil, folinic acid, and oxaliplatin in patients with advanced gastric cancer. J Clin Oncol. 2004 Feb 15;22(4):658-63. doi: 10.1200/JCO.2004.07.042. PMID 14966088
- [Background] Louvet C, Andre T, Tigaud JM, Gamelin E, Douillard JY, Brunet R, Francois E, Jacob JH, Levoir D, Taamma A, Rougier P, Cvitkovic E, de Gramont A. Phase II study of oxaliplatin, fluorouracil, and folinic acid in locally advanced or metastatic gastric cancer patients. J Clin Oncol. 2002 Dec 1;20(23):4543-8. doi: 10.1200/JCO.2002.02.021. PMID 12454110
- [Background] Diaz-Rubio E, Evans TR, Tabemero J, Cassidy J, Sastre J, Eatock M, Bisset D, Regueiro P, Baselga J. Capecitabine (Xeloda) in combination with oxaliplatin: a phase I, dose-escalation study in patients with advanced or metastatic solid tumors. Ann Oncol. 2002 Apr;13(4):558-65. doi: 10.1093/annonc/mdf065. PMID 12056706
- [Background] Cassidy J, Tabernero J, Twelves C, Brunet R, Butts C, Conroy T, Debraud F, Figer A, Grossmann J, Sawada N, Schoffski P, Sobrero A, Van Cutsem E, Diaz-Rubio E. XELOX (capecitabine plus oxaliplatin): active first-line therapy for patients with metastatic colorectal cancer. J Clin Oncol. 2004 Jun 1;22(11):2084-91. doi: 10.1200/JCO.2004.11.069. PMID 15169795
- [Background] Shields AF, Zalupski MM, Marshall JL, Meropol NJ. Treatment of advanced colorectal carcinoma with oxaliplatin and capecitabine: a phase II trial. Cancer. 2004 Feb 1;100(3):531-7. doi: 10.1002/cncr.11925. PMID 14745869
- [Background] de Gramont A, Figer A, Seymour M, Homerin M, Hmissi A, Cassidy J, Boni C, Cortes-Funes H, Cervantes A, Freyer G, Papamichael D, Le Bail N, Louvet C, Hendler D, de Braud F, Wilson C, Morvan F, Bonetti A. Leucovorin and fluorouracil with or without oxaliplatin as first-line treatment in advanced colorectal cancer. J Clin Oncol. 2000 Aug;18(16):2938-47. doi: 10.1200/JCO.2000.18.16.2938. PMID 10944126
- [Background] Sumpter, K., et al. Randomised, mulitcenter phase III study comparing capecitabine with fluorouracil and oxaliplatin with cisplatin in patients with advanced oesophagogastric cancer: confirmation of dose escalation. in Proc Am Soc Clin Onocol. 2003.
- [Background] Chong G, Cunningham D. Can cisplatin and infused 5-fluorouracil be replaced by oxaliplatin and capecitabine in the treatment of advanced oesophagogastric cancer? The REAL 2 trial. Clin Oncol (R Coll Radiol). 2005 Apr;17(2):79-80. doi: 10.1016/j.clon.2004.12.004. No abstract available. PMID 15830568
- [Background] Hurwitz H, Fehrenbacher L, Novotny W, Cartwright T, Hainsworth J, Heim W, Berlin J, Baron A, Griffing S, Holmgren E, Ferrara N, Fyfe G, Rogers B, Ross R, Kabbinavar F. Bevacizumab plus irinotecan, fluorouracil, and leucovorin for metastatic colorectal cancer. N Engl J Med. 2004 Jun 3;350(23):2335-42. doi: 10.1056/NEJMoa032691. PMID 15175435
- [Background] Giantonio, B., et al. High-dose bevacizumab in combination with FOLFOX4 improves survival in patients with previously treated advanced colorectal cancer: Results from the Eastern Cooperative Oncology Group (ECOG) study E3200. in Proc Am Soc Clin Oncol. 2005.
- [Background] Miller, K.D., et al. E2100: A randomized phase III trial of paclitaxel versus paclitaxel plus bevacizumab as first line threapy for locally recurrent or metastatic breast cancer. in American Society for Clinical Oncology. 2005. Orlando, FL.
- [Background] Shah, M.A., et al. A Multicenter Phase II Study of Irinotecan (CPT), Cisplatin (CIS), and Bevacizumab (BEV) in Patients with Unresectable or Metastatic Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma. in Proc Am Soc Clin Oncol. 2005.
- [Background] Goldberg, R.M., et al. N9741: oxaliplatin (Oxal) or CPT-11 + 5-fluorouracil (5FU)/leucovorin (LV) or oxal + CPT-11 in advanced colorectal cancer (CRC). Updated efficacy and quality of life (QOL) data from an intergroup study. in Proc Am Soc Clin Oncol. 2003.
- [Background] Takimoto CH, Remick SC, Sharma S, Mani S, Ramanathan RK, Doroshow J, Hamilton A, Mulkerin D, Graham M, Lockwood GF, Ivy P, Egorin M, Schuler B, Greenslade D, Goetz A, Knight R, Thomas R, Monahan BP, Dahut W, Grem JL; National Cancer Institute Organ Dysfunction Working Group Study. Dose-escalating and pharmacological study of oxaliplatin in adult cancer patients with impaired renal function: a National Cancer Institute Organ Dysfunction Working Group Study. J Clin Oncol. 2003 Jul 15;21(14):2664-72. doi: 10.1200/JCO.2003.11.015. PMID 12860942
- [Background] Xeloda Investigator Drug Brochure (Ro 09-1978), in Version 6. January 2002.
- [Background] Ishitsuka, H., T. Ishikawa, and Y. Fukase. Capecitabine and the dThdPase up-regulators IFN-gamma or taxol showed synergistic activity in human cancer xenografts. in Proc Am Assoc Cancer Res. 1996.
- [Background] Giantonio, B.J., et al. Incorporating angiogenesis inhibition with bevacizumab (anti-VEGF) into frontline chemotherapy with irinotecan (CPT-11), fluorouracil and leucovorin (FU/LV) for advanced colorectal cancer (advCRC): a toxicity analysis of ECOG study E2200. in Proc Am Soc Clin Oncol. 2002.
- [Background] Hochster, H., et al. Bevacizumab (B) with oxaliplatin (O)-based chemotherapy in the first-line therapy of metastatic colorectal cancer (mCRC): Preliminary results of the randomized ﾓTREE-2ﾔ trial. in Proc Am Soc Clin Oncol. 2005.
- [Background] Poon RT, Fan ST, Wong J. Clinical implications of circulating angiogenic factors in cancer patients. J Clin Oncol. 2001 Feb 15;19(4):1207-25. doi: 10.1200/JCO.2001.19.4.1207. PMID 11181687
- [Background] Lockhart AC, Braun RD, Yu D, Ross JR, Dewhirst MW, Klitzman B, Yuan F, Grichnik JM, Proia AD, Conway DA, Mann G, Hurwitz HI. A clinical model of dermal wound angiogenesis. Wound Repair Regen. 2003 Jul-Aug;11(4):306-13. doi: 10.1046/j.1524-475x.2003.11411.x. PMID 12846919
- [Background] Lockhart AC, Braun RD, Yu D, Ross JR, Dewhirst MW, Humphrey JS, Thompson S, Williams KM, Klitzman B, Yuan F, Grichnik JM, Proia AD, Conway DA, Hurwitz HI. Reduction of wound angiogenesis in patients treated with BMS-275291, a broad spectrum matrix metalloproteinase inhibitor. Clin Cancer Res. 2003 Feb;9(2):586-93. PMID 12576422
- [Background] Holden SN, Eckhardt SG, Basser R, de Boer R, Rischin D, Green M, Rosenthal MA, Wheeler C, Barge A, Hurwitz HI. Clinical evaluation of ZD6474, an orally active inhibitor of VEGF and EGF receptor signaling, in patients with solid, malignant tumors. Ann Oncol. 2005 Aug;16(8):1391-7. doi: 10.1093/annonc/mdi247. Epub 2005 May 19. PMID 15905307
- [Background] Chang HY, Sneddon JB, Alizadeh AA, Sood R, West RB, Montgomery K, Chi JT, van de Rijn M, Botstein D, Brown PO. Gene expression signature of fibroblast serum response predicts human cancer progression: similarities between tumors and wounds. PLoS Biol. 2004 Feb;2(2):E7. doi: 10.1371/journal.pbio.0020007. Epub 2004 Jan 13. PMID 14737219
- [Background] Hurwitz, H., et al. Wound healing/bleeding in metastatic colorectal cancer patients who undergo surgery during treatment with bevacizumab. in Proc Am Soc Clin Oncol. 2004.
- [Background] Scappaticci, F., et al. Analysis of wound healing and bleeding post-surgery in metastatic colorectal cancer patients treated with bevacizumab. in Proc Am Soc Clin Oncol. 2004.
- [Background] Gerber HP, Kowalski J, Sherman D, Eberhard DA, Ferrara N. Complete inhibition of rhabdomyosarcoma xenograft growth and neovascularization requires blockade of both tumor and host vascular endothelial growth factor. Cancer Res. 2000 Nov 15;60(22):6253-8. PMID 11103779
- [Background] Kim ES, Serur A, Huang J, Manley CA, McCrudden KW, Frischer JS, Soffer SZ, Ring L, New T, Zabski S, Rudge JS, Holash J, Yancopoulos GD, Kandel JJ, Yamashiro DJ. Potent VEGF blockade causes regression of coopted vessels in a model of neuroblastoma. Proc Natl Acad Sci U S A. 2002 Aug 20;99(17):11399-404. doi: 10.1073/pnas.172398399. Epub 2002 Aug 12. PMID 12177446
- [Background] Brookmeyer, R. and J.J. Crowley, A confidence interval for the median survival time. Biometrics, 1982. 38: p. 29-41.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 81 subjects consented, 21 were screen failures, 60 subjects were considered enrolled.
Groups:
- 1 - Capecitabine (Xeloda), Oxaliplatin and Bevacizumab (Avasti: capecitabine (Xeloda), oxaliplatin and bevacizumab (Avastin): Capecitabine will be administered orally at a twice daily dose of 850 mg/m2 (equivalent to a total daily dose of 1700 mg/m2) given days 1-14 of the three week cycle.
  Oxaliplatin will be administered at the dose of 130 mg/m2 given as a 2-hour intravenous infusion on day 1 of a three week cycle.
  Bevacizumab will be administered at a dose of 15 mg/kg given as a 30-90 minute intravenous infusion on day 1 of a three week cycle following the administration of oxaliplatin.
Period: Overall Study
Arm/Group | 1 - Capecitabine (Xeloda), Oxaliplatin and Bevacizumab (Avasti
Started | 60 (2 subjects signed the ICF, but were withdrawn from study prior to receiving any study drug)
Completed | 58
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Number of subjects receiving study drug
Groups:
- 1- Capecitabine (Xeloda), Oxaliplatin and Bevacizumab (Avastin: capecitabine (Xeloda), oxaliplatin and bevacizumab (Avastin): Capecitabine will be administered orally at a twice daily dose of 850 mg/m2 (equivalent to a total daily dose of 1700 mg/m2) given days 1-14 of the three week cycle.
  Oxaliplatin will be administered at the dose of 130 mg/m2 given as a 2-hour intravenous infusion on day 1 of a three week cycle.
  Bevacizumab will be administered at a dose of 15 mg/kg given as a 30-90 minute intravenous infusion on day 1 of a three week cycle following the administration of oxaliplatin.
Arm/Group | 1- Capecitabine (Xeloda), Oxaliplatin and Bevacizumab (Avastin
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 47

OUTCOME MEASURES:

1. Primary Outcome: Median Progression-Free Survival (PFS)
Description: Time in months from the start of study treatment to the date of first progression (PD) according to the RECIST criteria, or death due to any cause. PER RECIST, a PD is indicated when there is at least a 20% increase in the sum of the longest diameters from target lesions relative to the smallest sum recorded since treatment is initiated. Median PFS was estimated using a Kaplan-Meier curve, and is the time at which 50% of patients remain alive without disease progression.
Time Frame: 5 years from study start date
Population: All patients with at least one scheduled restaging who received treatment. However, an additional 3 patients who progressed before treatment are not included in this analysis.
Measure: Median (90% Confidence Interval); unit: survival time in months
Arm/Group | 1- Capecitabine (Xeloda), Oxaliplatin and Bevacizumab (Avastin
Number analyzed (Participants) | 49
survival time in months | 6.97 [6.41 to 8.15]

2. Secondary Outcome: To Assess the Safety and Tolerability of the Combination of Bevacizumab, Oxaliplatin and Capecitabine in Patients With Previously Untreated Metastatic Esophagogastric Adenocarcinoma
Description: Number of subjects who experienced an adverse event
Time Frame: Every 21 days
Measure: Number; unit: participants
Arm/Group | 1 - Capecitabine (Xeloda), Oxaliplatin and Bevacizumab (Avasti
Number analyzed (Participants) | 58
participants | 56

3. Secondary Outcome: Response Rate
Description: The proportion of patients for whom the best overall response is complete response (CR) or partial response (PR). A CR occurs when all lesions disappear; whereas, a PR is indicated when there is at least a 30% decrease in the sum of the longest diameters (LD) of the target lesion. A PD (progressive disese) occurs when there is at least a 20% increase in the sum of the LD relative to the smallest sum LD recorded since treatment is initiated. Disease is considered stable if there is no response and no PD. All patients were assigned a best response for inclusion in this calculation in accordance with the protocol.
Time Frame: Every 9 weeks for up to 1 year
Population: All eligible patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 1 - Capecitabine (Xeloda), Oxaliplatin and Bevacizumab (Avasti
Number analyzed (Participants) | 60
percentage of participants | 41.7 [29.1 to 55.1]

4. Secondary Outcome: Median Survival
Description: Time in months from the start of study treatment to date of death due to any cause. Median survival was estimated using a Kaplan-Meier curve and is the time point at which 50% of patients remain alive.
Time Frame: 5 years after study start date
Population: All patients who received treatment are included in the analysis population. However, 2 patients who never started treatment before leaving the study were excluded from this analysis of survival time.
Measure: Median (90% Confidence Interval); unit: survival time in months
Arm/Group | 1 - Capecitabine (Xeloda), Oxaliplatin and Bevacizumab (Avasti
Number analyzed (Participants) | 58
survival time in months | 10.51 [8.61 to 12.22]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from first dose of study drug until 30 days after last dose of study drug.
Arm/Group | 1 - Capecitabine (Xeloda), Oxaliplatin and Bevacizumab (Avasti
Serious Adverse Events (participants affected / at risk) | 33/58
Other Adverse Events (participants affected / at risk) | 56/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1 - Capecitabine (Xeloda), Oxaliplatin and Bevacizumab (Avasti (N=58)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Duodenal hemorrhage (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 2
Esophageal hemorrhage (Gastrointestinal disorders) | 1
Esophageal obstruction (Gastrointestinal disorders) | 1
Esophageal perforation (Gastrointestinal disorders) | 1
Gastric perforation (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 6
Death NOS (General disorders) | 1
Fatigue (General disorders) | 1
Pain (General disorders) | 3
Infections and infestations - Other, specify (Infections and infestations) | 3
Lung infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Anorexia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dysphasia (Nervous system disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Thromboembolic event (Vascular disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1 - Capecitabine (Xeloda), Oxaliplatin and Bevacizumab (Avasti (N=58)
Anemia (Blood and lymphatic system disorders) | 6
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 3
Sinus tachycardia (Cardiac disorders) | 1
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Blurred vision (Eye disorders) | 4
Eye disorders - Other, specify (Eye disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 7
Anal mucositis (Gastrointestinal disorders) | 3
Ascites (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 18
Diarrhea (Gastrointestinal disorders) | 26
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 5
Esophageal obstruction (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 6
Hemorrhoids (Gastrointestinal disorders) | 1
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 28
Oral pain (Gastrointestinal disorders) | 2
Rectal hemorrhage (Gastrointestinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 4
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 23
Chills (General disorders) | 1
Edema limbs (General disorders) | 4
Facial pain (General disorders) | 1
Fatigue (General disorders) | 28
Fever (General disorders) | 6
General disorders and administration site conditions - Other, specify (General disorders) | 3
Pain (General disorders) | 12
Hepatic failure (Hepatobiliary disorders) | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1
Allergic reaction (Immune system disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 6
Lung infection (Infections and infestations) | 1
Nail infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 4
Alkaline phosphatase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 5
Blood bilirubin increased (Investigations) | 4
CPK increased (Investigations) | 1
Investigations - Other, specify (Investigations) | 1
Neutrophil count decreased (Investigations) | 16
Platelet count decreased (Investigations) | 10
Weight loss (Investigations) | 10
White blood cell decreased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 24
Dehydration (Metabolism and nutrition disorders) | 6
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4
Buttock pain (Musculoskeletal and connective tissue disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 6
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Depressed level of consciousness (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 9
Dysgeusia (Nervous system disorders) | 9
Dysphasia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 4
Nervous system disorders - Other, specify (Nervous system disorders) | 5
Peripheral motor neuropathy (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 32
Syncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 2
Confusion (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 4
Personality change (Psychiatric disorders) | 1
Hemoglobinuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2
Urinary frequency (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 5
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 7
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Nail loss (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 17
Purpura (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 6
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 4
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 8
Hypotension (Vascular disorders) | 2
Thromboembolic event (Vascular disorders) | 4
Vascular disorders - Other, specify (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No